CLINICAL TRIAL: NCT06894199
Title: Work2Prevent Plus: Structural Intervention to Promote HIV Care in Black Sexual Minority Men
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); TaskForce Prevention & Community Services (Unknown); Chicago Black Gay Men's Caucus (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB22-0783; K08MH130253 (NIH)
Record Dates: First submitted 2025-03-03; First posted 2025-03-25 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Young Black sexual male: Participate in two day employment program
  Interventions: Other: The Work Shop
- Employment program facilitators: Lead or support the two day employment program
  Interventions: Other: The Work Shop

INTERVENTIONS:
Other: The Work Shop — Employment intervention consists of 2 days (about 5 hours each) of interactive educational content focused on a variety of topics.

SUMMARY:
The goal of this observational study is to learn about the pilot test of the employment program among young Black sexual minority men.

The main question it aims to answer is: What is the feasibility and acceptability of the employment program?

Young Black sexual minority male participants will attend the two day employment program and will complete four study surveys over the course of 13 months.

Employment program facilitators will complete a study survey and participate in a focus group over the course of 1 day.

DETAILED DESCRIPTION:
For this trial, we will recruit, screen, and enroll a sample of 120 young black sexual minority men from our networks of community-based organizations and LGBT-serving partners. Eligible participants will be pre-screened for enrollment by a University of Chicago study research staff/project manager. Next, the research staff will explain the scope of employment program and expectations of enrollees. Those interested in enrolling in the employment program and study will then be invited to an initial session of the employment program.

The overall employment program will consist of 2 days of workshop content focused on employment skills and the relationship between work and health.

Day One. Upon arrival, the program implementers and researchers will explain the employment program and purpose of the research study. University of Chiago research staff will complete informed consent procedures with participants prior to beginning the study baseline questionnaire and ensure that all participants are capable of consenting to participate. Participants will be asked to complete a release of information to access electronic medical records for the purposes of collecting measures of viral load and clinical care visit attendance at each time point.

Baseline (T1). Prior to the start of the first session, participants will be given an iPad tablet and headphones containing a 30-35 minute audio-computer assisted self-interview (ACASI) survey. Self-assessment measures, including: sociodemographic characteristics: age, race/ethnicity, income, incarceration history, and employment history; employment and housing: job seeking self-efficacy, average hours worked in a week (last 30 days), work motivation, job-seeking behavior, and homelessness (last 3 months); and clinical care: receipt of ART/PrEP prescription (past 4 months), visits for HIV/PrEP care (past 6 months), HIV/STI testing visits (past 6 months).

Day Two. Immediate-post program (T2). At the completion of the employment program on the second day, participants will complete a 25-30 minute ACASI survey assessing the feasibility, acceptability, and satisfaction with the employment program.

6-months (T3) and 12-months (T4) post-program. Participants will be contacted by study research staff to complete additional follow-up surveys via private phone conversation or independent completion online through the REDCap data collection platform. Follow-up surveys at 6 months and 12 months post-program will assess all variables addressed at T1.

ELIGIBILITY:
Inclusion Criteria:

* Identifying as male
* Having ever had sex with another man
* Being ages 18-29 years old
* Identifying as Black or African American OR
* Being ages 18 or older
* Participated in facilitation or administrative support for the program, "The Work Shop," at a partnering community-based organization

Exclusion Criteria:

- Participated in the preceding employment intervention, "Work2Prevent"

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Young black sexual male cohort will be selected from primary care clinics serving young sexual minority males; local gathering places and events for young sexual minority males, such as night clubs, House & Ball events, and other public places that serve the LGBTQ community (e.g., LGBTQ centers).
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-04-22 (Estimated)

PRIMARY OUTCOMES:
Acceptability of intervention | Post-Intervention, week 2
  Average score among participants of the Information Systems Success Model. The 16-item scale measures information quality, perceived usefulness, and overall satisfaction. Every item is scored on a 1-7 scale, with 1 being "Strongly Disagree" and 7 being "Strongly Agree". Responses are averaged to produce an overall ISSM score (1-7; higher scores indicate higher acceptability/satisfaction).
Satisfaction with intervention | Post-Intervention, week 2
  Average score among participants of the Information Systems Success Model. The 16-item scale measures information quality, perceived usefulness, and overall satisfaction. Every item is scored on a 1-7 scale, with 1 being "Strongly Disagree" and 7 being "Strongly Agree". Responses are averaged to produce an overall ISSM score (1-7; higher scores indicate higher acceptability/satisfaction).
Workshop feasibility | Immediately after the intervention
  Number of participants that complete at least two workshops
Missed sexual healthcare visits | Baseline, 6 months and 12 months
  Ratio of scheduled sexual healthcare visits to missed sexual healthcare visits in the past 6 months
Change in participants perceived ability and confident to perform job seeking activities | Baseline through 12 months
  Average change in score between baseline and 12 months on Job-Seeking Self-Efficacy scale on participants perceived ability and confidence to perform job seeking activities. The 12-item Job Seeking Self-Efficacy scale uses response values on a 1-10 score, with 1 being "Not at All Confident" and 10 being "Very Confident". Responses are averaged to yield a total score, with higher scores indicating higher self-efficacy. Change in JSS will be calculated by subtracting the JSS score at baseline (T1) from the JSS score at the 6- (T3) and 12-month follow-ups (T4) (-9 to +9; negative change indicates decreased self-efficacy, while positive change indicates increased self-efficacy).

SECONDARY OUTCOMES:
Change in hours worked per week | Baseline through 12 months
  Average change in number of reported hours worked each week between baseline and 12 months
Change in self-reported sexual risk behaviors | Baseline through 12 months
  Average change in self-reported sexual risk behaviors from baseline through 12 months. Sexual risk behaviors will be measured using 7 (8 for trans male participants) yes/no items assessing for engagement in the following behaviors during the past 6 months:
  1. Condomless anal intercourse (insertive)
  2. Condomless vaginal intercourse (insertive)
  3. Condomless anal intercourse (receptive)
  4. Condomless vaginal intercourse (receptive) - trans men only
  5. Intercourse while under the influence of alcohol
  6. Intercourse while under the influence of marijuana
  7. Intercourse while under the influence of stimulants
  8. Intercourse while under the influence of opioids Responses will be averaged at each assessment. Change in sexual risk behaviors will be calculated by subtracting the baseline value from follow-up (T3 and T4, respectively) values (range: -1 to +1; negative change indicates fewer sexual risk behaviors, while positive change indicates more sexual risk behaviors).

CONTACTS AND LOCATIONS:
Overall Officials: Darnell Motley, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
A dataset that has been deidentified will be uploaded to a research data repository at the end of the study. All collected IPD from participants in the trial will be included.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available 6 months after the primary paper from the study is published.
Access Criteria: Sharing criteria to be determined